CLINICAL TRIAL: NCT05632523
Title: Surveillance Pharmacologique et Immunitaire précoce après Conversion au Belatacept Chez Les Patients Ayant Subi Une Transplantation rénale : étude Pilote
Brief Title: Early Pharmacological and Immune Monitoring After Conversion to Belatacept in Renal Transplant Patients
Acronym: EPIMAC-BELA
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR210053
Record Dates: First submitted 2022-11-07; First posted 2022-11-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Renal Transplant; Conversion
Keywords: Blood sample; Urinary sample
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urinary
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adult patients with renal transplant: Conversion from anticalcineurin to belatacept
  Interventions: Other: Blood sample; Other: urinary sample

INTERVENTIONS:
Other: Blood sample — Blood samples are taken at each visit to the day hospital for a programmed belatacept perfusion
Other: urinary sample — Urinary samples are taken at each visit to the day hospital for a programmed belatacept perfusion

SUMMARY:
Single-center, prospective, translational, clinical-biological, multidisciplinary study

DETAILED DESCRIPTION:
All patients starting belatacept will be informed about non-interventional study and will be included unless they do not accept (non-opposition, consent is not required). Patients will be included and followed up during the 6 first months, i.e. 9 infusions. Blood samples (3 heparinized tubes of 7ml + 1 dry tube without separator gel of 5ml, i.e. 26ml maximum per sample) and urine samples will be harvested before each perfusions and in case of rejection. Clinical and biological data will be collected in an electronic CRF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Renal transplant patient
* Patient converted from an anticalcineurin to belatacept

Exclusion Criteria:

* Opposition to data processing
* Hemoglobin < 9g/dL
* Patient under judicial protection
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with renal transplant, converted from an anticalcineurin to belatacept at the Tours CHRU.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Lymphocyte subpopulations in blood before freezing | Day 0
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood before freezing | Day 14
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood before freezing | Day 28
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood before freezing | Day 42
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood before freezing | Month 2
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood before freezing | Month 3
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood before freezing | Month 4
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood before freezing | Month 5
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood before freezing | Month 6
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Day 0
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Day 14
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Day 28
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Day 42
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Month 2
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Month 3
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Month 4
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Month 5
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in blood after freezing | Month 6
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Day 0
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Day 14
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Day 28
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Day 42
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Month 2
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Month 3
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Month 4
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Month 5
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine before freezing. | Month 6
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Day 0
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Day 14
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Day 28
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Day 42
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Month 2
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Month 3
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Month 4
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Month 5
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry
Lymphocyte subpopulations in urine after freezing. | Month 6
  Variability in absolute counts and relative proportions immunological analyses in flow cytometry

SECONDARY OUTCOMES:
residual concentrations of belatacept | Day 0
  pharmacological analyses by mass spectrometry
residual concentrations of belatacept | Day 14
  pharmacological analyses by mass spectrometry
residual concentrations of belatacept | Day 28
  pharmacological analyses by mass spectrometry
residual concentrations of belatacept | Day 42
  pharmacological analyses by mass spectrometry
residual concentrations of belatacept | Month 2
  pharmacological analyses by mass spectrometry
residual concentrations of belatacept | Month 3
  pharmacological analyses by mass spectrometry
residual concentrations of belatacept | Month 4
  pharmacological analyses by mass spectrometry
residual concentrations of belatacept | Month 5
  pharmacological analyses by mass spectrometry
residual concentrations of belatacept | Month 6
  pharmacological analyses by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GATAULT, Principal Investigator — University Hospital, Tours
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided